CLINICAL TRIAL: NCT05162001
Title: Body Weight Response With Disulfiram in Humans. Concept Testing Study
Brief Title: Body Weight Response With Disulfiram in Humans
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Laboratorios Doctor Macías (Unknown)
Responsible Party: Principal Investigator, Alejandro E. Macias, Tenure professor, Universidad de Guanajuato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Disulfiram-01-2021
Record Dates: First submitted 2021-11-14; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Drug
Keywords: Obesity; Overweight; Obesity drug
MeSH Terms: conditions — Obesity; Overweight | interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disulfiram (Experimental): A group of adults with a body mass index bigger than 22, treated with disulfiram
  Interventions: Drug: Disulfiram 250 mg

INTERVENTIONS:
Drug: Disulfiram 250 mg — Disulfiram used qd during nine weeks to observe effects on body weight
  Other Names: Antabuse

SUMMARY:
Overweight and obesity due to food that exceeds the requirements is an increasingly common global problem. Lifestyle intervention and anorectic drugs result in minimal weight loss, which tends to be easily regained. In addition, drugs tend to have too many side effects and have had to be withdrawn from management schemes and even from the market. Disulfiram (Antabuse®️) is approved by the Food and Drug Administration against chronic alcohol addiction. In a mouse study, disulfiram prevented body weight gain and negated the adverse impact of an obesogenic diet on insulin; used properly it is a safe drug. Carrying out a testing-concept study with disulfiram will allow the establishment of guidelines on clinical studies focused on its use as an adjunct in the reduction and control of body weight.

DETAILED DESCRIPTION:
BACKGROUND Overweight and obesity due to food that exceeds the requirements is an increasingly common global problem. It is considered one of the great public health challenges because it leads to the so-called "metabolic syndrome" and its associates such as diabetes mellitus, hypertension and non-alcoholic steatohepatitis. In 2016, more than 1.9 billion adults aged 18 and over were overweight, of which more than 650 million were obese. It is estimated that if nothing is done, by 2030 about half of the world's adult population will have obesity.

Multiple paths have been taken to reverse overweight and obesity, with poor results. Lifestyle intervention and anorectic drugs result in minimal weight loss, which tends to be easily regained. In addition, drugs tend to have too many side effects and have had to be withdrawn from management schemes and even from the market. In Mexico, for example, there are aberrant commercial presentations of drugs that include anorectics, benzodiazepines, thyroid hormones, and atropinic drugs in a single capsule. Bariatric surgery is more effective, but it is an extreme solution that is reserved for patients with morbid obesity and it is associated with its own postoperative morbidity and mortality. Therefore, it is urgent to have new therapeutic elements that help to lose weight effectively and permanently; otherwise, there is no way out of this global problem.

One of the most attractive study targets for developing anti-overweight drugs is the dynamics of body fat. Adipose tissue is not inert, but participates in the control of appetite, glucose homeostasis, insulin sensitivity, and body temperature. White adipose tissue (WAT) stores important energy reserves. Brown adipose tissue (BAT) is an important site of thermo genesis, essential for maintaining body temperature regulated by mitochondrial uncoupling protein 1 (UCP-1), which is activated by exposure to cold. The WAT can acquire characteristics of the BAT thanks to a "browning", which is the appearance of brown fat within deposits of white fat; this improves thermo genesis, increases energy expenditure, and potentially reduces obesity. This browning and its metabolic changes have been achieved in mice with the use of digoxin, thanks to the inhibition of the Interleukin-17 (IL-17) axis.

Disulfiram (Antabuse®) is approved by the Food and Drug Administration against chronic alcohol addiction. In a mouse study, disulfiram prevented body weight gain and prevented the adverse impact of an obesogenic diet on insulin; furthermore, it reverted established diet-induced obesity and metabolic dysfunctions, apparently due to a reduction in feeding efficiency and an increase in energy expenditure; Also in mice treated with disulfiram, loss of fatty tissue, reduction of steatohepatitis and reduction of hyperplasia of the pancreatic islets have been observed, apparently due to the promotion of autophagy. Given the potent anti-obesogenic effects in rodents, clinical reassignment of disulfiram could represent a new strategy to treat obesity and its metabolic comorbidities. In the present study, the investigators proposed a proof-of-concept design to observe the safety of the use of disulfiram in adults with a body mass index greater than 22, as well as the eventual response of body weight and serum metabolic indicators.

JUSTIFICATION

The various strategies used to achieve control and reduction in body weight of overweight and obese subjects have shown little effectiveness. Achieving control in body weight and even a significant decrease in it, is associated with positive outcomes for the health of patients. There is in vivo evidence regarding the use of disulfiram in obese mice where a significant decrease in weight and an improvement in metabolic aspects were achieved. Disulfiram is a drug approved for use in the control of alcohol addiction; used properly it is safe. Carrying out a proof-of-concept study with disulfiram will allow the establishment of guidelines on clinical studies focused on its use as an adjunct in the reduction and control of body weight.

PROBLEM STATEMENT

Given the failure of various strategies to control and decrease body weight in overweight or obese patients, there is in vivo evidence regarding the use of disulfiram as a regulator of body weight in mice. Therefore, it is proposed to carry out a study in ten human volunteers to answer the following question:

Is the use of disulfiram for 9 weeks safe and does it significantly affect body weight?

HYPOTHESIS

H0: The use of disulfiram for 9 weeks does not significantly decrease body weight.

Hi: Using disulfiram for 9 weeks significantly decreases body weight.

OBJECTIVES General objective. To determine if the use of disulfiram for 9 weeks significantly decreases body weight.

Particular objectives.

1. Describe the anthropometric and clinical characteristics of the participants at the beginning and end of the study.
2. Compare the anthropometric and clinical characteristics of the participants at the beginning and at the end of the study.
3. Describe the effect of disulfiram on the body weight of the participants.
4. Determine if there is a significant variation in the body weight of the participants.
5. Determine if there are side effects of disulfiram in volunteers, determined by clinical or laboratory parameters.

MATERIAL AND METHODS

Type of study: Clinical trial for proof of concept.

Study design: Non-comparative prospective longitudinal experimental study.

Population sample Sample size calculation: A minimum sample size of ten volunteers was determined by considering an alpha probability of 0.05, a statistical power of 0.80 and a difference of 3% of body weight at the end of the study. The calculation was made based on the following formula: n = (Zα / 2 + Zβ) 2 * 2 * σ2 / d2, where Zα / 2 is the critical value of the normal distribution in α / 2 (for example, for a 95% confidence level, α is 0.05 and the critical value is 1.96), Zβ is the critical value of the normal distribution in β (for example, for an 80% power, β is 0.2 and the critical value is 0.84), σ2 is the population variance and d is the difference to detect.

After the inclusion of two volunteers, a preliminary analysis will be done to determine if the study should continue, based on side effects, safety concerns, or significant change in body weight.

Recruitment instructions On recruitment, the research subject will be given clear instructions and instructed to follow their usual diet, without making an effort to lose weight. Disulfiram will be administered at a dose of 500 mg per day for one week, to continue at 250 mg per day for 9 weeks. Participants will be warned of the danger of alcohol in relation to the intake of disulfiram, as it can cause serious reactions. Participants should not take metronidazole or paraldehyde, or any food or product that contains alcohol (including mouthwashes, cough medicines, wine or vinegar for cooking, certain desserts and chocolates, as well as any that the subject identifies). Participants will not drink alcohol in any amount while taking disulfiram and for 14 days after taking the last dose.

As an extra precaution, the volunteer will be asked to avoid the use of products that could lead to skin absorption of small amounts of alcohol or vinegar, such as after-shave products, colognes, perfumes, antiperspirants, skin products, antiseptics, astringents, hair dyes and others. Participants will be instructed to check the label to see if any food or medicine contains alcohol. Also, participants will avoid contact with non-consumable products that may contain alcohol, such as paint thinners, solvents, dyes, lacquers and others.

Variables

Age, gender, height, initial weight, initial body mass index in Kg/m2 will be determined. Subsequently, daily weight in the morning fasting for 8 hours or more, with light underwear, at the same time of day and on the same clinical scale (Tanita 585f, Tokyo, Japan), which have a precision of +/- 100 g.

Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Hematic cytology, Erythrocyte sedimentation rate, C-reactive protein, Glucose, Creatinine, Total bilirubins, Alanine transaminase (ALT), aspartate transaminase (AST), Cholesterol, triglycerides, High-density lipoprotein (HDL) cholesterol, Low-density lipoprotein (LDL) cholesterol (calculated), general urine test.

ANALYSIS The variables will be recorded on a capture sheet and their analysis will be carried out according to their nature. For the descriptive analysis of the quantitative variables, means and their standard deviation or medians and their inter-quartile range (Q1 to Q3) will be reported, depending on whether the data is normal or not in its distribution; on the other hand, for the qualitative variables, percentages, proportions or rates will be reported, as appropriate. The normality in the distribution of the data will be carried out using the Shapiro-Wilk test.

The comparative analysis of the quantitative variables will be carried out using parametric or non-parametric inferential tests, depending on the nature of the distribution of the variables. The change in body weight will be determined in absolute and relative values (Kg). To consider that there is a significant change, a difference of at least 3% in weight relative to 9 weeks is established. This analysis will be performed using the paired t-test or the Wilcoxon signed rank test. Changes in qualitative variables will be made using the McNemar test. A value of p <0.05 will be considered significant. The data analysis will be carried out using the statistical package NCSS(r) statistical Software (2018). (12.0.2. NCSS(r), LLC. Kaysville, Utah, USA, ncss.com/software/ncss).

ETHICAL ASPECTS The project was submitted for approval to the Research and Research Ethics Committee of the ISSSTE hospital, Leon Mexico. This research protocol is based on the Mexican General Health Law, and corresponds to a study with greater than minimal risk (Chapter I, Article 17, section III), complies with the provisions of Articles 13, 14, 16, 19, 20 , 21,22, in relation to studies in humans. In the same way, it adheres to the Helsinki declaration adopted by the 64th World Medical Assembly, Fortaleza, Brazil (2013), and refers to the recommendations to guide health personnel in biomedical research with human beings, in addition to following the international codes and statutes active to date for proper practice in the field of clinical research. This investigation will be guided under the principles of beneficence, non-maleficence, justice and autonomy indicated in the Belmont report.

Study staff will follow good clinical practice recommendations. The research center where all the data will be recorded (Laboratorios Doctor Macias), will be audited at least once per month by personnel of the "Instituto de Seguridad y Servicios Sociales para los Trabajadores del Estado" (ISSSTE) hospital assigned to the research and ethics areas.

The privacy of patients and the confidentiality of the data that allow their identification will be protected. Patients must voluntarily accept their participation and sign a letter of consent.

All adverse events and serious adverse events will be reported classifying them into 3 groups: not related to study procedures, probably related to study procedures and directly related to study procedures.

All members of the study staff declare that they have no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* 18 to 65 years old
* height >160 cm
* fast weight >65 Kg
* Body Mass Index (BMI) >22.

Exclusion Criteria:

* Diabetes
* vascular diseases
* liver diseases
* renal failure
* cancer
* chronic obstructive pulmonary disease (COPD)
* alcohol, drugs or tobacco addiction
* convulsive diseases
* hypothyroidism
* tuberculosis or chronic debilitating diseases
* use of statins or other lipid lowering drugs
* anticoagulants drugs
* herbal remedies.
* For women 18 to 50 years old, pregnancy should ruled out with a proper test before recruiting and anti conceptive measures must be started in case of active sexual life during all the time of the study and 2 additional weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Body weight change | nine weeks
  Daily weight in the morning fasting for 8 hours or more, with light underwear, at the same time of day and on the same clinical scale (Tanita 585f, Tokyo, Japan), which have a precision of +/- 100 g.

SECONDARY OUTCOMES:
Changes in hematic cytology | nine weeks
  Laboratory test within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Hematic cytology. Units of measurement: cells by mm^3
Changes in Erythrocyte sedimentation rate. | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Erythrocyte sedimentation rate. Unit of measurement: mm/hour
Changes in C-reactive protein. | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: C-reactive protein. Unit of measurement: mg/L
Changes in glucose | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Glucose. Unit of measurement: mg/dL
Changes in creatinine. | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Creatinine. Unit of measurement: mg/dL
Changes in total bilirubins. | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: total bilirubins. Unit of measurement: mg/dL.
Changes in Alanine- Aminotransferase. | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Alanine-Aminotransferase Unit of measurement: IU/L
Changes in Aspartate-aminotransferase | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Aspartate-aminotransferase. Unit of measurement: IU/L
Changes in cholesterol | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Cholesterol. Unit of measurement: mg/dL
Changes in triglycerides | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: Triglycerides. Unit of measurement: mg/dL
Changes in HDL cholesterol | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: HDL cholesterol. Unit of measurement: mg/dL
Changes in LDL cholesterol | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: LDL cholesterol. Unit of measurement: mg/dL
Changes in General urine test | nine weeks
  Laboratory tests within 72 hours before the start of the study, as well as 7 days and the last day of treatment and four weeks after the end of treatment. Blood tests with a minimum fasting of 8 h: General urine test. Unit of measurement: positive/negative

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro E Macias, MD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- University of Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
It will be shared with other researchers as solicited, as long as the individual participants agree.

REFERENCES:
- [Background] Hall KD, Kahan S. Maintenance of Lost Weight and Long-Term Management of Obesity. Med Clin North Am. 2018 Jan;102(1):183-197. doi: 10.1016/j.mcna.2017.08.012. PMID 29156185
- [Result] Chouchani ET, Kazak L, Spiegelman BM. New Advances in Adaptive Thermogenesis: UCP1 and Beyond. Cell Metab. 2019 Jan 8;29(1):27-37. doi: 10.1016/j.cmet.2018.11.002. Epub 2018 Nov 29. PMID 30503034
- [Result] Seale P, Conroe HM, Estall J, Kajimura S, Frontini A, Ishibashi J, Cohen P, Cinti S, Spiegelman BM. Prdm16 determines the thermogenic program of subcutaneous white adipose tissue in mice. J Clin Invest. 2011 Jan;121(1):96-105. doi: 10.1172/JCI44271. Epub 2010 Dec 1. PMID 21123942
- [Result] Teijeiro A, Garrido A, Ferre A, Perna C, Djouder N. Inhibition of the IL-17A axis in adipocytes suppresses diet-induced obesity and metabolic disorders in mice. Nat Metab. 2021 Apr;3(4):496-512. doi: 10.1038/s42255-021-00371-1. Epub 2021 Apr 15. PMID 33859430
- [Result] Bernier M, Mitchell SJ, Wahl D, Diaz A, Singh A, Seo W, Wang M, Ali A, Kaiser T, Price NL, Aon MA, Kim EY, Petr MA, Cai H, Warren A, Di Germanio C, Di Francesco A, Fishbein K, Guiterrez V, Harney D, Koay YC, Mach J, Enamorado IN, Pulpitel T, Wang Y, Zhang J, Zhang L, Spencer RG, Becker KG, Egan JM, Lakatta EG, O'Sullivan J, Larance M, LeCouteur DG, Cogger VC, Gao B, Fernandez-Hernando C, Cuervo AM, de Cabo R. Disulfiram Treatment Normalizes Body Weight in Obese Mice. Cell Metab. 2020 Aug 4;32(2):203-214.e4. doi: 10.1016/j.cmet.2020.04.019. Epub 2020 May 14. PMID 32413333
- [Result] Bernier M, Harney D, Koay YC, Diaz A, Singh A, Wahl D, Pulpitel T, Ali A, Guiterrez V, Mitchell SJ, Kim EY, Mach J, Price NL, Aon MA, LeCouteur DG, Cogger VC, Fernandez-Hernando C, O'Sullivan J, Larance M, Cuervo AM, de Cabo R. Elucidating the mechanisms by which disulfiram protects against obesity and metabolic syndrome. NPJ Aging Mech Dis. 2020 Jul 21;6:8. doi: 10.1038/s41514-020-0046-6. eCollection 2020. PMID 32714562